CLINICAL TRIAL: NCT06279845
Title: A Multicenter Prospective Clinical Cohort Study on the Pathogen Spectrum of Hepatic Virus-caused Cirrhosis Complicated With Infection
Brief Title: A Clinical Cohort Study on the Pathogen Spectrum of Hepatic Virus-caused Cirrhosis Complicated With Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Zhejiang University (Other)
Collaborators: Beijing Ditan Hospital (Other); Beijing YouAn Hospital (Other); Huashan Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Jiajia Chen, Chief Physician of the First Affiliated Hospital,Zhejiang University School of Medicine, Zhejiang University
Other Study IDs: 2023YFC2308802-02
Record Dates: First submitted 2024-02-18; First posted 2024-02-28 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Liver Cirrhosis
Keywords: Hepatic virus-caused cirrhosis; Infection; Pathogen spectrum; Cohort study
MeSH Terms: conditions — Liver Cirrhosis; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — According to the characteristics of infection, take blood or body fluids from the corresponding infected site.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to expound the population and characteristics of pathogenic microorganisms with co-infection, draw the pedigree of pathogenic microorganisms, and evaluate its influence on disease outcome in patients with hepatic virus-caused cirrhosis. The main questions it aims to answer are:

* Describe the populations and characteristics of pathogenic microorganisms responsible for co-infections in patients with hepatic virus-caused cirrhosis.
* Map the spectrum of pathogenic microorganisms, and evaluate their impact on disease regression.

DETAILED DESCRIPTION:
Cirrhosis is a chronic progressive disease caused by different etiological factors and characterized by diffuse hepatocellular degeneration and necrosis, abnormal regeneration of hepatocytes, intrahepatic neovascularization, massive proliferation of hepatic fibrotic tissues, and pseudofollicular formation. The number of patients with liver disease in China is about 300 million, and the number of deaths from cirrhosis accounts for 11% of the global deaths from cirrhosis. Its etiology is diverse, and hepatitis due to hepatophilic virus infection is still the main cause in China. A recent study by scholars on 11861 patients hospitalized for the first time due to liver cirrhosis in 50 hospitals in China showed that among the causes of liver cirrhosis in China, HBV infection accounted for 71.15% and HCV infection accounted for 8.12%. About two-thirds of patients with cirrhosis and extrahepatic organ failure suffer from sepsis. Infections increase the risk of death in patients with cirrhosis, and reports have shown that these patients are hospitalized for twice as long as patients without cirrhotic sepsis and have a hospital mortality rate of up to 50%. This study focuses on the impact of secondary infections on the clinical prognosis of cirrhosis, and proposes to establish a prospective, multicenter clinical cohort of secondary infections in cirrhosis, map infection pathogens, correlate the characteristics of the underlying immune status with the pathogen profiles of secondary infections, and set up an early warning system of secondary infection surveillance, with the aim of early prevention and early recognition of secondary infections, and improvement of prognosis for patients with liver cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients with viral hepatitis cirrhosis agreed to participate in the study and signed an informed consent form;
2. Any gender and age between 18-70 years old;
3. HBsAg positivity lasting more than 6 months;
4. have clinical manifestations of hepatic decompensation and portal hypertension, laboratory test results, liver imaging or endoscopy and other comprehensive diagnosis of definite cirrhosis.

Exclusion Criteria:

1. Patients with other non-hepatophilic causes of cirrhosis;
2. Patients who, in the opinion of the investigator, are not suitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatic virus-caused cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Secondary infection in patients at 4 weeks | 4 weeks
  Site of infection, pathogen results such as blood or body fluid pathogen cultures or Next-generation sequencing(NGS) results.
quick SEPSIS RELATED ORGAN FAILURE ASSESSMENT(qSOFA) at 4 weeks | 4 weeks
  qSOFA consists of 3 items: altered state of consciousness, systolic blood pressure ≤ 100 mmHg, and respiratory rate ≥ 22 respirations/min. 2 or more items, i.e., a qSOFA score of ≥ 2, are considered to be suspicious for sepsis.Higher qSOFA scores are associated with a higher risk of patient death.

SECONDARY OUTCOMES:
Survival rate | 12 weeks
  12-week survival in infected patients with viral hepatitis cirrhosis

CONTACTS AND LOCATIONS:
Overall Officials: Jiajia Chen, Principal Investigator — Zhejiang University